CLINICAL TRIAL: NCT02716844
Title: The Effect Of The Clinical Pilates Exercises On Kinesiophobia, And Other Symptoms Related to Osteoporosis
Brief Title: Effect Of Exercises On Kinesiophobia, And Other Symptoms Related to Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Sevim Öksüz, Senior Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LUT11/16,B:30.2.HAC.0.20.05.04
Record Dates: First submitted 2016-03-03; First posted 2016-03-23 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Clinic Pilates Exercise; Kinesiophobia; Pain
MeSH Terms: conditions — Osteoporosis; Kinesiophobia; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Group, (Experimental): Clinical Pilates exercise were given for 6 weeks, 3 days in a week
  Interventions: Other: Exercise
- Control Group (No Intervention): Nothing given to control group, told to continue their normal life for 6 weeks.

INTERVENTIONS:
Other: Exercise — Clinical Pilates exercise were given for 6 weeks, 3 days in a week
  Arms: Exercise Group,

SUMMARY:
Aim: Investigating the effects of Clinical Pilates Exercise on kinesiophobia, pain, functional status and quality of life of the patients diagnosed with osteoporosis.

Method: 47 patients were assessed and randomly divided into 2 groups. Exercise group patients joined exercise program regularly that was held 3 times a week, 1 hour a day, during 6 weeks with physiotherapist. Control group patients continued their normal daily lives without any exercise. After 7 patients quit the study for various reasons, 40 women with primary osteoporosis (control group n=20, exercise group n= 20), completed the study and were assessed at the beginning and at the end of 6 weeks. As assesment' measurements Tampa Kinesiophobia Scale (TKS), Visual Analog Scale (VAS), Short Form McGill (SF-McGill), Pain Disability Index (PDI), Oswestry Disability Index (ODI), Berg Balance Test (BBT), Timed Up- Go Test (TUG), Chair Sit-Stand Test (CSST), Chair Sit and Reach Test (CSRT), Back Scratch Test (BST), Quality of life Questionnaire European Foundation for Osteoporosis (QUALEFFO-41), Hospital Anxiety and Depression Scale (HADS), Satisfaction with Life Scale (SLS) and Health Assesment Questionnaire (HAQ) were performed.

ELIGIBILITY:
Inclusion Criteria:

* Woman diagnosed with osteoporosis between the ages 50-75 within the last year

Exclusion Criteria

* History of fractures
* Joint replacements or fixation of the joints at the lower extremities or the spine
* Any neurological or muscle diseases
* Inability to continuously attend the exercise program
* Any secondary diseases resulting in decreased mobility or functional status
* Visual, hearing or mental problems that could prevent communication

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the level of fear and avoidance associated with movement assessed using the Tampa Kinesiophobia Scale at 6 weeks | At the beginning and at the end of 6 weeks
  40 osteoporosis patients filled Tampa Kinesiophobia Scale at the beginning and at the end of 6 weeks in order to measure the level of fear and avoidance associated with movement. If an individual receives a high score, according to the scale, this result indicates a high level of kinesiophobia . It has not a specific unit. There is not an adverse events in this test.

SECONDARY OUTCOMES:
Change in the level of pain intensity in the morning assessed using Visual Analogue Scale (VAS) at 6 weeks. | At the beginning and at the end of 6 weeks
  VAS is an horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current pain intensity. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks and recorded in centiemeters (cm).
Change in the level of pain intensity during activity assessed using Visual Analogue Scale (VAS) at 6 weeks. | At the beginning and at the end of 6 weeks
  VAS is an horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current pain intensity. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks and recorded in centiemeters (cm).
Change in the level of pain intensity at rest assessed using Visual Analogue Scale (VAS) at 6 weeks. | At the beginning and at the end of 6 weeks
  VAS is an horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current pain intensity. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks and recorded in centiemeters (cm).
Change in the level of experienced pain assessed with using Short Form - McGill Pain Questionnaire (SF-McGill) | At the beginning and at the end of 6 weeks
  Short Form - McGill Pain Questionnaire (SF-McGill) provides a multidimensional evaluation of the experienced pain. Patients' pain descriptions (SF-McGill S), experienced pain level during study (Sf-McGill VAS) and total pain intensity measured via a 6-point Likert- Type Scale (SF-McGill L) was recorded.
Change in the level of influence of patients' general pain intensity on their daily life activities and functionality assessed using Pain Disability Index (PDI). | At the beginning and at the end of 6 weeks
  Pain Disability Index (PDI) (score out of 70) is a questionnaire filled by the patients.
Change in the level of influence of patients' low back pain intensity on their daily life activities and functionality assessed using Oswestry Low Back Pain Disability Scale (ODI) | At the beginning and at the end of 6 weeks
  Oswestry Low Back Pain Disability Scale (ODI)(score out of 70) is a questionnaire filled by the patients .
Change in the level of functional balance assessed using Berg Balance Test (BBT). | At the beginning and at the end of 6 weeks
  Berg Balance Test (BBT)(score out of 56) evaluates postural control mechanism and dynamic and static balance while doing functional activities in adult population. This test was assessed by the physiotherapist.
Change in the level of functional balance assessed using The Timed Up and Go Test (TUG). | At the beginning and at the end of 6 weeks
  The Timed Up and Go Test (TUG) assesses the functional balance and mobility of subjects. Patients stands up upon therapist's command walks 3 meters, turns around, walks back to the chair and sits down. The performance is repeated by the patience 3 times and the shortest performance time is recorded in seconds (sec).
Change in the level of lower extremity proximal muscle's strength and endurance assessed using Chair Sit and Stand Test (CSST) at 6 weeks. | At the beginning and at the end of 6 weeks
  In Chair Sit and Stand Test (CSST), number of sitting-standing repetitions in 30 sec. was recorded by the physiotherapist.
Change in the level of functional flexibility of lower extremity assessed using Chair Sit and Stand Test (CSST) at 6 weeks. | At the beginning and at the end of 6 weeks
  assesses the functional flexibility of the lower extremity in adult (23). Participant sits on the edge of a chair. One foot must remain flat on the floor. The other leg is extended forward with the knee straight, heel on the floor, and ankle bent at 90°. Patients place one hand on top of the other with tips of the middle fingers even. Patients keep the knee straight, and hold the reach for 2 seconds. If the fingertips touch the toes then the score is zero (0). If they do not touch, measure the distance between the fingers and the toes (a negative score/-), if they overlap, measure by how much (a positive score/+) and recorded in cm.
Change in the level of functional flexibility of upper extremity assessed using Back Scratch Test (BST) at 6 weeks. | At the beginning and at the end of 6 weeks
  Back Scratch Test (BST)(cm) evaluates the functional flexibility of the patient's upper extremity. Patients are asked to rotate their shoulder externally with palms facing their back. Their hand fingers extend while trying to reach the lowest point, the other arm internally rotates while trying to reach the highest point. Patients are asked their fingertips to be closer to each other. If finger tips do not touch each other, the distance between them is recorded in cm assumed as a negative score, if the fingertips touch each other, then the score is assumed as zero. If they overlap, it is recorded in cm taking as positive score. Three repetitions are performed consecutively and the best score was recorded.
Change in the level of quality of life assessed using Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) at 6 weeks | At the beginning and at the end of 6 weeks
  A. Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) examine the five dimensions of health such as pain, physical functioning, social activities, general health assessment and mental function of patients with osteoporosis. Quality of Life Questionnaire of the European Foundation for Osteoporosis (QUALEFFO-41) was filled by the patients and score was calculated as percentage (%).
Change in the level of anxiety and depression assessed using Hospital Anxiety And Depression Scale (HADS) at 6 weeks | At the beginning and at the end of 6 weeks
  This scale was filled by the patients. It has no special units. The elevation of the total score indicates the increased anxiety and depression levels (score out of 42).
Change in the level of chronic functional impairment assessed using Health Assessment Questionnaire (HAQ) at 6 weeks | At the beginning and at the end of 6 weeks
  Health Assessment Questionnaire (HAQ) (score out of 24) is commonly used for evaluating the patients' chronic functional impairment caused by rheumatic diseases. This questionnaire was filled by the patients and it has no special units.
Change in the level of life satisfaction assessed using Satisfaction with Life Scale (SLS) at 6 weeks | At the beginning and at the end of 6 weeks
  This scale (score out of 35) was filled by the patients. It has no special units.

IPD SHARING:
Plan to Share IPD: Undecided